CLINICAL TRIAL: NCT05222347
Title: Evaluation of the Immunomodulatory and Preventive Effects of Olive Leaf Tea Against COVID-19
Brief Title: Immunomodulatory and Preventive Effects of Olive Leaf Tea Against COVID-19
Status: Completed | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Collaborators: Albayraklar Foundation (Unknown)
Responsible Party: Sponsor
Other Study IDs: SBUSAH GETAT 2020-011
Record Dates: First submitted 2022-02-01; First posted 2022-02-03 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2022-02

CONDITIONS: Immunomodulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Comparison of biochemical parameters of OLT drinkers: Compared biochemical parameters of OLT smokers and nonsmokers
  Interventions: Dietary Supplement: Olive Leaf Tea
- Comparison of biochemical parameters of OLT nondrinkers: Compared biochemical parameters of OLT smokers and nonsmokers
  Interventions: Dietary Supplement: Olive Leaf Tea

INTERVENTIONS:
Dietary Supplement: Olive Leaf Tea — Olive-leaf tea (OLT) is widely used in the traditional medicine in the Mediterranean region. Due to the high concentration of phenolic compounds, of which most abundant is oleuropein, interest in olive leaf has increased recently [22, 23]. The components of the olive leaves are known for their immune-modulatory, anti-inflammatory, antioxidant, hypoglycemic, antihypertensive, antimicrobial, and anti-atherosclerotic effects [24, 25]. Although its antiviral mechanism of action is not fully known, many studies have been conducted on the antiviral effects of olive leaf extract .

SUMMARY:
During the Coronavirus Disease-2019 (COVID-19) pandemic, in addition to the current measures, boosting the immune system seems to be one of preventive measures that can be taken against COVID-19 infection. Various natural agents have been recommended to boost the immune system. The aim of this study was to investigate the possible immunomodulatory and preventive effects of Olive Leaf Tea (OLT) drinking with regards to COVID-19 infection. The study was conducted among 249 workers in a tractor factory where OLT was served. Of the 249 workers, 168 of them were OLT drinkers and 81 were not OLT drinkers. Drinking at least one cup of OLT per day for a minimum of one month was the inclusion criteria used in the study. The workers with a history of infection or vaccination of COVID-19 were excluded. Lymphocyte subsets, IL2, INF-gamma, specific IgM, and IgG levels were analyzed in all the study subjects. The results showed higher values of CD3-/CD16/56 (NK) cells, CD3+/CD16/56 (NKT) cells, total NK (NK+NKT) cells, and serum IFN-gamma and IL-2 levels in OLT drinkers as compared to the nondrinkers. These immune changes are indicative of immune defense mechanisms. Although all the OLT drinkers and non-drinkers reported no history of COVID-19, specific COVID-19 IgG levels were found positive in 60% of OLT drinkers and 38% OLT non-drinkers. There were significant negative correlations between age and NK cells, number of cigarettes smoked and NK cells, number of cigarettes smoked and TNK; and there were positive correlations between OLT drinking frequency and TNF-alpha, IL-2 and IFN-gamma. Also, serum creatinine levels in OLT non-drinkers were found significantly higher than in the OLT drinkers. In conclusion, drinking OLT may contribute fighting against COVID-19 by boosting the innate immune system.

DETAILED DESCRIPTION:
Coronavirus Disease-2019 (COVID-19) is caused by severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2). It emerged out of China in late 2019 and rapidly led to a pandemic in early 2020. As the mutations of the virus continue to increase, the pandemic has become difficult to control and no specific treatment has been proven to be effective.

According to the European Centre for Disease Prevention and Control (ECDC), until a safe and effective vaccine is available, non-pharmaceutical tools are accepted as the most effective public health interventions against COVID-19. World Health Organization (WHO) states that in addition to public health and social measures, it is also beneficial for individuals to maintain a balanced diet, stay well hydrated, exercise regularly and sleep well.

It is now clear that there is a close interaction between the COVID-19 and the immune system of an individual resulting in diverse clinical manifestations of the disease. While some patients present severe complications, some individuals remain asymptomatic. Weakened immunity is responsible for most COVID-19 deaths, therefore, elderly people with chronic diseases are considered at high risk from COVID-19.

As soon as SARS-CoV-2 binds to angiotensin converting enzyme 2 (ACE2) receptors and releases viral RNA for replication, both the innate and adaptive immune responses are triggered. Natural killer (NK) cells are innate effector lymphocytes that play a critical role in the first line of defense against tumor cells and viral infections. They are essential in the early immune response against viral infections, mainly through the clearance of virus-infected cells. Human NK cells, CD3-CD56+ NK, represent an average of 15% of peripheral blood and they can be subdivided based on the relative expression of the surface markers CD16 and CD56. Additionally, in chronic viral infections, CD56-CD16+ NK cells are expanded and seems to represent an exhausted/anergic subset of NK cells. Through several mechanisms, NK cells provide exocytosis of perforin and granzyme causing lysis of the infected cell, Fas ligand-mediated induction of apoptosis, and antibody-dependent cellular cytotoxicity (ADCC), while having an essential role as immunomodulatory cells that bridge the innate and adaptive immune responses. Natural killer T cells (NKT) are cells that express a semi-invariant T cell receptor (TCR). Crucial cytokines for the cytotoxic activity of NK and NKT cells are IL-2 and INF-gamma, and these cytokines enhance the killing properties and proliferation of these cells. Both IL-2 and IFN-gamma secretions are induced in a healthy young individual while this effect decreases in the elderly.

Immune system boosting nutrition may play a role to lower the risk of infections by inhibiting virus replication, promoting virus clearance, inducing tissue repair, and triggering a prolonged adaptive immune response against viruses. Besides, certain medicinal plants are known for their antiviral bioactivities and immune boosting capacity. Some herbs have immunomodulatory potential and can be applied as a preventive medicine to combat COVID-19. Olive-leaf tea (OLT) is widely used in the traditional medicine in the Mediterranean region. Due to the high concentration of phenolic compounds, of which most abundant is oleuropein, interest in olive leaf has increased recently. The components of the olive leaves are known for their immune-modulatory, anti-inflammatory, antioxidant, hypoglycemic, antihypertensive, antimicrobial, and anti-atherosclerotic effects. Although its antiviral mechanism of action is not fully known, many studies have been conducted on the antiviral effects of olive leaf extract . However, studies on the protective or immune system strengthening effect of olive leaf extract against viral diseases are limited. There is only one available in vitro study that shows olive leaf extract alters the immune response by increasing the number of CD8 + and NK cells and IFN-gamma. The aim of this study is to investigate the possible immunomodulatory and preventive effects of OLT against COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Health male subjects aged between 20-60

Exclusion Criteria:

-Those who drank less than three cups of OLT a day were excluded from the study.

Ages: 20 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: workers at the Tumosan Konya tractor factory
Sampling Method: Probability Sample
Enrollment: 249 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-03-04 (Actual); Study Completion 2021-09-05 (Actual)

PRIMARY OUTCOMES:
Olive Leaf Tea increase immune force and prevent COVID-19 infection | One year

CONTACTS AND LOCATIONS:
Overall Officials: Eray M. Guler, Assoc. Prof., Principal Investigator — University of Health Sciences Turkey, Hamidiye School of Medicine, Dept. of Medical Biochemistry; Arzu Irban, Professor, Principal Investigator — University of Health Sciences Turkey, Hamidiye School of Medicine, Department of Anesthesiology,; Bayram Kiran, Professor, Principal Investigator — Kastamonu University, Faculty of Engineering and Architecture, Dept. of Genetics and Bioengineering
Locations (1):
- Tumosan Konya Tractor Factory, Konya, Selcuklu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
We will not use the participants data

REFERENCES:
- [Derived] Kocyigit A, Guler EM, Irban A, Kiran B, Atayoglu AT. Assessment of Association Between the Potential Immunomodulatory Activity and Drinking Olive Leaf Tea in the Coronavirus Disease-2019 Pandemic: An Observational Study. J Integr Complement Med. 2022 Dec;28(12):940-947. doi: 10.1089/jicm.2022.0554. Epub 2022 Sep 16. PMID 36112183